CLINICAL TRIAL: NCT02351271
Title: A Single Centre Randomized Eye Study to Compare the Performance and Safety of Femtosecond Laser-assisted Cataract Procedures With Conventional Ultrasound-assisted Cataract Surgery
Brief Title: Cataract Surgery: Femto LDV Z8 Versus Conventional
Acronym: COMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL5940-0996
Record Dates: First submitted 2015-01-16; First posted 2015-01-30 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femto LDV Z8 (Experimental): Femtosecond laser-assisted cataract pre-treatment: Capsulotomy and lens fragmentation, followed by ultrasound phacoemulsification
  Interventions: Device: Femto LDV Z8
- Manual capsulorhexis&lens fragmentation (Active Comparator): The Conventional group acts as a control group with conventional capsulorhexis and ultrasound phacoemulsification
  Interventions: Device: Manual capsulorhexis&lens fragmentation

INTERVENTIONS:
Device: Femto LDV Z8 — Femtosecond laser-assisted cataract pre-treatment: Capsulotomy and lens fragmentation, followed by ultrasound phacoemulsification
  Other Names: Treatment A
  Arms: Femto LDV Z8
Device: Manual capsulorhexis&lens fragmentation — Control treatment where the capsulorhexis is performed manually and the lens fragmentation is performed by the stop and chop technique with the phaco emulsification device
  Other Names: Treatment B
  Arms: Manual capsulorhexis&lens fragmentation

SUMMARY:
The aim of the study is to demonstrate the performance and safety of the Femtosecond laser-assisted anterior capsulotomy and lens fragmentation on human eyes using the FEMTO LDV Z8 compared to conventional technique in cataract surgery.

DETAILED DESCRIPTION:
Cataract Surgery according to conventional procedure, with the exception of two steps (Capsulotomy and Lens Fragmentation) which are performed with a Femtosecond Laser in the study group. Used equipment for measurements is the same for both groups and in line with the normal equipment used for the conventional cataract treatment (group A) Cataract surgery will be performed conventionally, this means the capsulorhexis will be performed manually by a hook, and the lens extraction will be done by phacoemulsification. (group B)

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo cataract extraction by phacoemulsification with primary intraocular lens Implantation
* Able to co-operate with the docking system for the femtosecond laser
* Clear corneal media
* 50 years of age or older
* Willing and able to return for scheduled follow-up examinations

Exclusion Criteria:

* Minimal and maximal K-values of the central 3mm zone that differ by more than 5D on a keratometric map of the cornea
* Maximum K-value that exceeds 58D
* Minimal K-value of less than 37D
* Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light
* Poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Manifest Glaucoma+OHT (ocular hypertension), pseudoexfoliation
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye
* Known sensitivity to planned concomitant medications
* History of lens or zonular instability
* Keratoconus or keratectasia
* Immune compromised or diagnosis of connective tissue disease, clinically sign. atopic disease, insulin dependent diabetes mellitus, autoimmune diseases, ocular herpes zoster or simplex, endocrine diseases, lupus, RA, collagenosis and other acute or chronic illnesses that increases the risk to the subject or confounds the outcomes of this study, in the opinion of the study PI.
* Anterior chamber depth (ACD) < 1.5 mm or ACD > 4.8 mm as measured from the corneal endothelium.
* Extensive corneal scarring
* Developmental disability or cognitive impairment (would preclude adequate comprehension of the Informed Consent (IC) form and/or the ability to record the study measurements)
* Concurrent participation in another ophthalmological clinical study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Pajic, MD, PhD, Principal Investigator — Augenzentrum ORASIS AG

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Femto LDV Z8: Femtosecond laser-assisted cataract pre-treatment: Capsulotomy and lens fragmentation, followed by ultrasound phacoemulsification
  Femto LDV Z8: Femtosecond laser-assisted cataract pre-treatment: Capsulotomy and lens fragmentation, followed by ultrasound phacoemulsification
  33 males (48.5%) and 35 females (51.5%) in the FLACS group
- Manual Capsulorhexis&Lens Fragmentation: The Conventional group acts as a control group with conventional capsulorhexis and ultrasound phacoemulsification
  Manual capsulorhexis&lens fragmentation: Control treatment where the capsulorhexis is performed manually and the lens fragmentation is performed by the stop and chop technique with the phaco emulsification device
  25 (40.3%) males and 37 females (59.7%) in the manual group
Period: Overall Study
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation
Started | 68 | 62
Completed | 68 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation | Total
Number analyzed (Participants) | 68 | 62 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 60 | 57 | 117
Age, Continuous [Mean (Full Range); unit: years] | 70.4 [50 to 83] | 69.6 [50 to 85] | 70 [50 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 33 | 25 | 58
Region of Enrollment [Number; unit: participants]
  Switzerland | 68 | 62 | 130

OUTCOME MEASURES:

1. Primary Outcome: Effective Phaco Time (EPT)
Description: Effective Phacoemulsification Time (EPT): EPT for eyes receiving Intervention A being statistically same or lower than EPT for eyes receiving Intervention B at p<0.05 will be considered positive for superior efficacy of application of FEMTO LDV Z8 over the manual procedure
  Effective Phaco Time is a unit. It is commonly understood in the area of cataract surgery to be the standard way to describe phaco energy during a procedure over different manufactured phaco devices.
  Effective phaco time is the total phaco time at 100 percent phaco power. It can be less than the total foot-pedal time. Less EPT indicates proportionately less energy delivered to the eye thereby reducing the side effects of phaco power.
Time Frame: day of surgery
Population: effective phaco time
Measure: Mean (Standard Deviation); unit: EPT
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation
Number analyzed (Participants) | 68 | 62
EPT | 1.48 (1.8) | 2.3 (2.41)

2. Secondary Outcome: Ease of Phacoemulsification
Description: Ease of phacoemulsification was performed as a subjective observation by the surgeon. Four classifications were possible: easy - phacoemulsification was fast and uncomplicated; 'slight resistance' - phacoemulsification encountered some difficulty; 'resistance noted' - phacoemulsification was somewhat complex; 'difficult' - phacoemulsification was difficult and complex to complete.
Time Frame: during surgery
Population: Participants were classified as 'easy' or as 'slight resistance' in terms of ease of phacoemulsification.
Measure: Count of Participants; unit: Participants
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation
Number analyzed (Participants) | 68 | 62
Participants
  Classification - easy | 66 | 59
  Classification - slight resistance | 2 | 3

3. Secondary Outcome: Number of Participants With Complete Treatment Pattern
Description: Completeness of capsulotomy is a subjective metric given by the surgeon. Measurements were scaled into the following four categories: 1: complete treatment pattern; 2: micro-adhesion; 3: incomplete treatment pattern; 4: complete pattern but not continuous. "Complete treatment pattern" is considered the best result, "micro adhesion" indicates a minor but manageable problem, "incomplete treatment pattern" indicates a treatable, but more complex suboptimal outcome and "complete treatment but discontinuous pattern" indicates the treatable but suboptimal outcome.
Time Frame: during surgery
Population: In all cases, the capsulotomy was categorized as a complete treatment pattern
Measure: Count of Participants; unit: Participants
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation
Number analyzed (Participants) | 68 | 62
Participants | 68 | 62

4. Other Pre Specified Outcome: Number of Participants With Reported Complications
Description: Safety will be assessed by evaluating observed and/or reported device and non-device related Adverse Events and/or Adverse Device Effects between treatment intervention groups A and B. No serious adverse events were reported. One AE in the femto group and two in the manual group were reported.
Time Frame: during follow-up after 1 and 12 days, 4, 8 and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation
Number analyzed (Participants) | 68 | 62
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: one year and 3 months
Description: AE and SAE defined same as clinicaltrials.gov. As both interventions are limited to the anterior segment of the eye which is a contained anatomical space, deaths due to the intervention of either study group are considered to be zero. However, for the purpose of this study, all AE, SAE and deaths will be monitored.
Arm/Group | Femto LDV Z8 | Manual Capsulorhexis&Lens Fragmentation
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/62
Other Adverse Events (participants affected / at risk) | 1/68 | 2/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Femto LDV Z8 (N=68) | Manual Capsulorhexis&Lens Fragmentation (N=62)
Transient IOP rise (Eye disorders) | 1 (1) | 0 (0) — Intraocular pressure
herpes zoster (Eye disorders) | 0 (0) | 1 (1)
postoperative edema of the optic disk (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less